CLINICAL TRIAL: NCT00095667
Title: A Phase 2 Study of GW572016 in Hormone Naive Recurrent or Metastatic Hormone Sensitive Prostate Cancer
Brief Title: Lapatinib in Treating Patients With Recurrent or Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03178; PHL-030; CDR394173; N01CM62203 (NIH)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Lapatinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Phase II trial to study the effectiveness of lapatinib in treating patients who have recurrent or metastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the antitumor activity of GW572016 in hormone naïve, recurrent and/or metastatic hormone sensitive prostate cancer using PSA response rate.

SECONDARY OBJECTIVES:

I. To estimate objective tumor response in patients with measurable disease. II. To determine the duration of PSA response, rate and duration of stable disease, progression-free, median and overall survival rates of GW572016 in recurrent and/or metastatic prostate cancer.

III. To document the safety and tolerability of GW572016 in these patient populations.

TERTIARY OBJECTIVES:

I. To investigate if differences in baseline levels of EGFR and/or erbB2 expression, and receptor phosphorylation status in tumor specimens predict outcome to therapy.

II. To investigate if the inhibitory effects of GW572016 on EGFR and/or erbB2 pathway activation in tumor specimens correlates with clinical outcome.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for this study within 11.7 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed prostate cancer that is recurrent after local therapy, and/or metastatic carcinoma confirmed to be of prostate origin
* Patients must have recurrent and/or metastatic disease that is progressive and not amenable to surgery or curative radiotherapy; progressive disease is defined as:

  * Three consecutive rising PSAs, at least 4 weeks apart with an absolute increase of at least 0.5
  * PSA doubling time of less than one year
  * PSA > 2.0
* For recurrent disease following local therapy (surgery/radiation), prior neoadjuvant or adjuvant hormones are allowed if completed more than a year prior to study entry; for metastatic disease, no prior medical therapy (hormonal, corticosteroid, chemotherapy) is allowed
* Life expectancy of greater than 12 weeks
* ECOG performance status 0,1, or 2
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan; note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution
* Must be willing and able to undergo tumor biopsy once before (if no previous specimen available) and once during investigational therapy if there are lesions accessible for biopsy for correlative studies; in cases where there is a medical contraindication to tumor biopsy, exception may be granted only upon discussion with the principal investigator
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of GW572016 will be determined following review of their use by the principal investigator
* Patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring INR
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Able to swallow and retain oral medication

Exclusion Criteria:

* Prior treatment:

  * Patients who have had prior chemotherapy for prostate cancer
  * Patients who have been on androgen ablative therapies within the last year
  * Patients receiving radiotherapy to the prostate less than 6 weeks prior to study entry
  * Patients who have had prior treatment with EGFR targeting therapies
  * Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy
* Patients with a history of other active malignancy in the past 5 years (with the exception of adequately treated non-melanomatous skin cancers) are excluded
* History of allergic reactions attributed to compounds of similar chemical or biological composition to GW572016
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with cardiac ejection fraction, not within the institutional range of normal as measured by echocardiogram or MUGA scan at baseline
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Concomitant requirement for medication classified as CYP3A4 inducer or inhibitor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
PSA response rate defined as at least a 50% fall in PSA from baseline confirmed by a second PSA 4 weeks later | Up to 3 years

SECONDARY OUTCOMES:
Objective tumor response | Up to 3 years
  Potential association between variables will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon tests may be substituted if necessary. Ninety-five percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Duration of PSA response | Up to 3 years
  Potential association between variables will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon tests may be substituted if necessary. Ninety-five percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Rate and duration of stable disease | From the start of the treatment until the criteria for progression are met, assessed up to 3 years
  Potential association between variables will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon tests may be substituted if necessary. Ninety-five percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Progression-free survival | From start of treatment to time criteria are met for disease progression, assessed up to 3 years
  Will be computed using the Kaplan-Meier method.
Overall survival | Up to 3 years
  Will be computed using the Kaplan-Meier method.
Safety and tolerability assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 3 years
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.

CONTACTS AND LOCATIONS:
Overall Officials: John Trachtenberg, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada